CLINICAL TRIAL: NCT06427525
Title: The Effect of Mobile Application Supported Health Promotion Program on Obesity, Physical Activity and Stress Levels of Adolescents
Brief Title: The Effect of Mobile Application Supported Health Promotion Program on Obesity of Adolescents
Acronym: obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cumali Yıldızdal, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Mobile Application Health
Record Dates: First submitted 2023-10-07; First posted 2024-05-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Adolescents; Mobile Application; School Health; Physical Activity; Nutrition Disorder, Child
MeSH Terms: conditions — Motor Activity; Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): mobile application at preventing overweight and obesity in childhood
  Interventions: Other: Mobile application-based adolecent obesity education
- Control group (No Intervention): health education

INTERVENTIONS:
Other: Mobile application-based adolecent obesity education — Mobile application-based adolecent obesity education
  Arms: Intervention group

SUMMARY:
The aim of the study is to evaluate the effectiveness of the Child Obesity Program (COP), which is a school-based, parent-based, weight management program aimed mobile application at preventing overweight and obesity in childhood.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of the Child Obesity Program (COP), which is a school-based, parent-based, weight management program aimed mobile application at preventing overweight and obesity in childhood. The program aims to provide children with positive health behaviors, gain cognitive and behavioral skills that will enable them to increase their knowledge of physical activity, nutrition and stress management.

ELIGIBILITY:
Inclusion Criteria:

Obesity Adolescents, smartphone internet, 10-16 years old

Exclusion Criteria:

non-obese child, 17 years old

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Healthy Lifestyle Behaviors Scale | 1 month
  higher scores mean a better

CONTACTS AND LOCATIONS:
Overall Officials: Cumali Yıldızdal, phd student, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Florance Nightingale Nursing Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No